CLINICAL TRIAL: NCT01222065
Title: Polarization Sensitive Retinal Tomography for Glaucoma Diagnosis
Acronym: PSOCT
Status: Completed | Type: Observational
Sponsor: Courtney Frazier Swaney (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Courtney Frazier Swaney, Office of Sponsored Projects, University of Texas at Austin
Organization: University of Texas at Austin (Other)
Other Study IDs: 2007-04-0101; R01EY016462 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Glaucoma
Keywords: Glaucoma; Neurotubules; Birefringence; Retinal Nerve Fiber Layer (RNFL)
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glaucoma/Normal: Two groups will be studies: patients with glaucomatous visual field loss and age and gender matched normal patients without visual field loss

SUMMARY:
The proposed human clinical studies have three main objectives:

1. To determine reproducibility of peripapillary birefringence maps and identify features that measure the health of the RNFL.
2. To determine the normal variation in the birefringence maps with age.
3. To develop and test a classifier for glaucoma based on the birefringence maps using a case-control clinical trial.

This study is a case-control study intended to optimize feature selection for a future multi-center blinded study. The proposed clinical study does not measure conversion from normal to glaucoma.

DETAILED DESCRIPTION:
This study evaluates RNFL Birefringence in normal and glaucoma human subjects: The primate experimental glaucoma study will characterize the spatial and temporal dynamics of RNFL birefringence during glaucoma progression and establish an initial feature set and classifier for a case-control clinical study. The case-control clinical study will refine the initial feature set and classifier and use ROC analysis to test sensitivity and specificity of the feature set and classifier for discriminating between normal and glaucomatous human eyes. The feature set and classifier formulated in the case-control clinical study is a prerequisite for planning a large-scale longitudinal study. A large-scale longitudinal study to compare different approaches for detecting early glaucoma is outside the scope of the proposed research. Moreover, considering the large number of subjects required for statistical significance when the conversion rate from ocular hypertensive to glaucoma is low (<10%/year), a longitudinal study is best performed in a multi-institution clinical trial over several years.

ELIGIBILITY:
Inclusion Criteria: patient age between 40 and 80, visual acuity score of 20/40 or better; spherical refraction within ± 5 diopters, cylinder refraction within ± 3 diopters, ability to cooperate with study procedures and personnel and to perform tests reliably. Case-control assignment for the human clinical trials is based on medical and ocular history and on a comprehensive eye examination (including intraocular pressure history, standard disc photography and Humphrey-Zeiss 24-2 visual field test) by a glaucoma specialist.

-

Exclusion Criteria: discernable anomaly of the anterior chamber, uveitis, significant opacification of the cornea or crystalline lens, eyes with secondary glaucoma, eyes with pigmentary or pseudoexfoliation glaucoma, concurrent active eye disease in the study eye that may affect intraocular pressure or its measurement, patients on kidney dialysis, eyes with proliferative or severe nonproliferative retinopathy, retinal detachment, retinitis pigmentosa, or other significant retinopathy, eyes with field loss attributed to a non-glaucoma condition, dilated pupil diameter less than 4mm, and visual fields < 20 degrees.

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 45 normal volunteers and 40 glaucoma patients (known visual field defects)with equal sex distribution between the ages of 40 and 80 will be recruited for this study by H. Grady Rylander, M.D. at The Eye Institute of Austin and grouped by age into the following categories: 40-49, 50-59, 60-69, 70-79. Every effort will be made to equalize the number of patients in each age category and to recruit volunteers representing the race distribution in our community. Maps of RNFLT, phase retardation, and RNFL birefringence will be acquired from individuals within each age category.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity/specificity of PSOCT to classify glaucoma vs. non-glaucoma | The time frame to assess the effectiveness of the diagnostic algorithm is 1 year
  Features from RNFL phase retardation and birefringence maps will be combined into a diagnostic algorithm to differentiate glaucoma vs. non-glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Henry G Rylander, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- Eye Institute of Austin, Austin, Texas, United States

REFERENCES:
- [Result] Park J, Kemp NJ, Rylander HG 3rd, Milner TE. Complex polarization ratio to determine polarization properties of anisotropic tissue using polarization-sensitive optical coherence tomography. Opt Express. 2009 Aug 3;17(16):13402-17. doi: 10.1364/oe.17.013402. PMID 19654746
- [Result] Pocock GM, Aranibar RG, Kemp NJ, Specht CS, Markey MK, Rylander HG 3rd. The relationship between retinal ganglion cell axon constituents and retinal nerve fiber layer birefringence in the primate. Invest Ophthalmol Vis Sci. 2009 Nov;50(11):5238-46. doi: 10.1167/iovs.08-3263. Epub 2009 Jun 3. PMID 19494208
- [Result] Liu S, Paranjape AS, Elmaanaoui B, Dewelle J, Rylander HG 3rd, Markey MK, Milner TE. Quality assessment for spectral domain optical coherence tomography (OCT) images. Proc SPIE Int Soc Opt Eng. 2009;7171:71710X. doi: 10.1117/12.809404. PMID 20431701
- See also: BME website with links to faculty — http://www.bme.utexas.edu